CLINICAL TRIAL: NCT04583085
Title: Interplay of miRNA-146a and miRNA-126 in Chronic Periodontitis Patients With Coronary Artery Disease
Status: Completed | Type: Observational
Sponsor: Meenakshi Ammal Dental College and Hospital (Other)
Responsible Party: Principal Investigator, Dr.Jaideep Mahendra, Professor, Director of PG education, Meenakshi Ammal Dental College and Hospital
Other Study IDs: MADC/IRB-XXVI/2018/415
Record Dates: First submitted 2020-10-03; First posted 2020-10-12 (Actual); Last update posted 2020-10-14 (Actual); Status verified 2020-10

CONDITIONS: Chronic Periodontitis; Coronary Artery Disease; miRNA
Keywords: Chronic Periodontitis; coronary artery disease; microRNA 146a; microRNA 126; plaque samples; biomarkers
MeSH Terms: conditions — Chronic Periodontitis; Coronary Artery Disease

STUDY DESIGN:
Observational Model: Other | Time Perspective: Other
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- CP + CHD group: This was further divided into CP + CHDa (Subgingival plaque) and CP + CHDb (Coronary plaque) based on the nature of plaque collected.
- CP group: 25 patients with chronic periodontitis who were systemically healthy were selected
- HP group: 25 patients who were systemically and periodontally healthy, were considered as HP group.

SUMMARY:
The role of micro-RNAs in chronic periodontitis associated with CAD is still in an incipient stage needs to be explored further. The investigators attempt to quantify and compare the levels of micro-RNA 146a and micro-RNA 126 in subgingival as well as coronary plaque samples obtained from patients diagnosed with chronic periodontitis with and without coronary artery disease.

DETAILED DESCRIPTION:
The role of micro-RNAs in chronic periodontitis associated with CAD is still in an incipient stage needs to be explored further. The investigators attempt to quantify and compare the levels of micro-RNA 146a and micro-RNA 126 in subgingival as well as coronary plaque samples obtained from patients diagnosed with chronic periodontitis with and without coronary artery disease.

Seventy-five participants were selected and grouped into 3 categories; 25 patients diagnosed with chronic periodontitis and coronary artery disease: CP + CAD group; 25 patients diagnosed with chronic periodontitis alone: CP group; and 25 systemically and periodontally healthy controls (HP). Demographic variables, periodontal parameters, cardiac parameters, blood pressure were obtained. miRNA-146a and miRNA126 levels were assessed in subgingival plaque (SP) samples from all the three groups. Within CP+CAD group, SP samples of CP+CADa were compared with coronary plaques samples (CP) of CP+CADb while the patient underwent CABG.

ELIGIBILITY:
Inclusion criteria:

* Patients volunteering for the investigation.
* Patients between the age group of 30-70 years
* Presence of ≥ 15 natural teeth.

Exclusion criteria:

* Patients associated with systemic diseases such as lung disorders, renal disease, liver disease, type I, type II-diabetes mellitus, HIV infection, rheumatoid arthritis, allergy or any malignancy.
* Under treatment with antibiotics, immunosuppressive drugs such as corticosteroids, within 6 months.
* Pregnant women and female patients were excluded because of the altered oral flora due to hormonal changes
* Smoking and other tobacco usage habits
* Patients who underwent periodontal treatment within 6 months.

Ages: 30 Years to 70 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Only male patients in the age group of 30-70 years were included. Females were excluded due to hormonal changes or pregnancy that may alter the oral flora
Study Population: Male subjects within 30-70 years of age were selected for the study
Sampling Method: Non-Probability Sample
Enrollment: 75 (Actual)
Dates: Start 2018-11-01 (Actual); Primary Completion 2019-12-01 (Actual); Study Completion 2019-12-31 (Actual)

PRIMARY OUTCOMES:
micro-RNA 146-a expression in Chronic periodontitis patients with and without coronary heart disease. | 10 months
  microRNA 146-a expression was present in the chronic periodontitis subjects with coronary heart disease
Levels of micro-RNA 126 in chronic periodontitis patients with and without coronary heart disease | 10 months
  microRNA 126 expression was present in chronic periodontitis subjects with coronary heart disease

CONTACTS AND LOCATIONS:
Locations (1):
- Meenakshi Ammal Dental college, Chennai, Tamil Nadu, India

IPD SHARING:
Plan to Share IPD: No